CLINICAL TRIAL: NCT00446212
Title: Dreaming and EEG Changes During Anaesthesia Maintained With Propofol or Desflurane
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2006.125
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Anaesthesia
Keywords: anaesthesia; propofol; desflurane; dreaming; electroencephalography
MeSH Terms: interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Propofol based anaesthetic maintenance with propofol effect-site steered target-controlled infusion, in addition to fentanyl and non-opioid analgesics
  Interventions: Drug: Propofol
- 2 (Active Comparator): Desflurane based anaesthetic maintenance with manually controlled administration in 100% oxygen in addition to fentanyl and non-opioid analgesics
  Interventions: Drug: desflurane

INTERVENTIONS:
Drug: Propofol — target controlled infusion of propofol
  Arms: 1
Drug: desflurane — Anaesthetic maintenance with desflurane
  Arms: 2

SUMMARY:
We hypothesise that patients who receive propofol for maintenance of anaesthesia will report dreaming more often when they emerge from anaesthesia than patients who receive desflurane for maintenance of anaesthesia.

DETAILED DESCRIPTION:
Patients commonly report that they have been dreaming when they emerge from anaesthesia. Data from observational studies and small randomised trials suggests that reports of dreaming are more commonly made after anaesthesia maintained with propofol than anaesthesia maintained with inhaled anaesthetic agents. We propose to randomise 300 healthy patients to receive a standardised general anaesthetic for surgery that includes either propofol or desflurane for maintenance. We will measure the raw and processed electroencephalogram during and after anaesthesia and interview patients about dreaming as soon as they emerge from anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Age between 18 and 50 years
* Presenting for elective surgery under general anaesthesia

Exclusion Criteria:

* Inadequate English language comprehension
* Major drug abuse problem

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Incidence of dreaming reported by patients interviewed immediately on emergence from anaesthesia using a standardised questionnaire | recovery room stay

CONTACTS AND LOCATIONS:
Overall Officials: Kate Leslie, MD, Principal Investigator — Melbourne Health
Locations (4):
- Australia (3):
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - King Edward Memorial Hospital for Women, Subiaco, Western Australia
- Waikato Hospital, Hamilton, New Zealand

REFERENCES:
- [Derived] Liang Z, Wang Y, Ren Y, Li D, Voss L, Sleigh J, Li X. Detection of burst suppression patterns in EEG using recurrence rate. ScientificWorldJournal. 2014;2014:295070. doi: 10.1155/2014/295070. Epub 2014 Apr 17. PMID 24883378
- [Derived] Leslie K, Sleigh J, Paech MJ, Voss L, Lim CW, Sleigh C. Dreaming and electroencephalographic changes during anesthesia maintained with propofol or desflurane. Anesthesiology. 2009 Sep;111(3):547-55. doi: 10.1097/ALN.0b013e3181adf768. PMID 19672164